CLINICAL TRIAL: NCT07125365
Title: UK Islet Autoantibody Registry
Acronym: UKIAb Registry
Status: Recruiting | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: Cardiff University (Other); University of Edinburgh (Other); University of Cambridge (Other); University of Dundee (Other); University of Birmingham (Other); Imperial College London (Other); University of Bristol (Other); King's College London (Other); Oxford University Hospitals NHS Trust (Other); University of Exeter (Other)
Responsible Party: Sponsor
Other Study IDs: PID:18612; IRAS Project ID: 347853 (Other: IRAS); REC reference: 25/SC/0089 (Other: Health Research Authority)
Record Dates: First submitted 2025-07-08; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-07

CONDITIONS: Type 1 Diabetes (T1D); Registry; Pre-diabetes; Screening
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Glucose Intolerance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- UKIAb: Children and adults aged 6 months - 70 years, positive for ≥ 1 islet autoantibody (IAb)

SUMMARY:
Type 1 diabetes (T1D) is a life-long condition where the immune system destroys part of the body (the pancreas) which makes the chemical, insulin. Insulin is needed to control blood sugar levels. Treatment involves life-long insulin replacement by injection or insulin pump.

Previous research has shown that the development of T1D occurs through different stages. This starts with a phase where there are no symptoms, which can last months or years, before symptoms of T1D develop and a person becomes unwell. The risk of developing T1D increases with presence of markers in the blood called islet autoantibodies. The risk of developing T1D increases with presence of markers in the blood called islet autoantibodies (IAb). Children with two or more IAb have an 80-90% chance of developing T1D within 15 years. It is almost certain that they will develop the condition in their lifetime. Children with only one IAb have a much lower risk of developing T1D (around 15%). Less is understood about the natural history of being IAb positive in adults, and the investigators hope this study will help them understand more.

The aim of the research is to understand what it is like to live with being at risk of T1D, what information and support people need, and whether they use NHS services more than others, for example due to being anxious about developing T1D. The investigators will work with the public and patient involvement group using information from the research and, with the charity Diabetes UK, to create a policy statement about the type of care that is needed to support these individuals.

To be able to do this research, tbhe investigators need first to recruit these rare individuals into one single registry of children, young people and adults who have islet autoantibodies in their blood. This will also allow the invetigators to collect data from individuals in the registry to compare this to data from other countries, to help understand why people progress from being islet autoantibody positive to requiring insulin in the UK.

People entering the registry will also be told if a drug is licensed in the UK to help delay T1D onset. Participants can also consent to be contacted about any research studies, which are testing drugs or interventions to prevent or delay the start of T1D.

DETAILED DESCRIPTION:
BACKGROUND AND RATIONALE Type 1 diabetes can be identified in the pre-clinical phase Understanding of the natural history of Type 1 diabetes (T1D) has made it possible to diagnose children, young people and adults (CYPA) in the preclinical phase. The presence of ≥ 2 Islet autoantibodies (IAb) in serum, to 4 different proteins (insulin, Glutamic Acid Decarboxylase (GADA), insulinoma-2-associated autoantibodies (IA-2A), and/or zinc transporter 8 autoantibodies (ZnT8A) identifies individuals who will develop T1D. The latency period before clinical diagnosis can last months or years, with individuals with ≥2 IAb moving between stage 1 (normoglycaemia), stage 2 (dysglycaemia) to stage 3 (hyperglycaemia), or clinical disease.

Data from combined longitudinal cohorts shows that ≥ 2 IAb in children predicts that stage 3 T1D will develop in over 80% over the next 15 years, and near 100% over a lifetime, whereas only around 10-15% children with a single IAb progress to insulin requirement. Individuals may therefore live for many years with the knowledge they may develop T1D .

Potential benefits of early identification of T1D Identifying T1D before symptoms develop has several potential advantages, including reducing presentation with life-threatening diabetic ketoacidosis (DKA) and its associated morbidity, and potentially reducing the psychological trauma at diagnosis which some families liken to 'post-traumatic distress' . Reducing DKA and hospitalisations can also reduce associated health care costs. Screening identifies individuals suitable for trials to prevent or delay T1D. Therapies are now being trialled in stage 2 T1D, for example, the ATG prevention trial 'STOP-T1D'.

Concerns about screening Informing someone that they have positive IAb may cause psychological stress. For example, the Fr1da study, which has now tested > 170,000 children for IAb, found that informing parents of their child's positive IAb result induced stress (assessed by the Patient Health Questionnaire-9); this stress declined after 12 months of follow up. Within the registry, the investigators have recourse to the advice of a senior clinical psychologist, who can provide signposting support for individuals identified through the registry, if psychological concerns arise.

Screening initiatives Until recently, screening strategies have focussed on first-degree relatives (FDR) of individuals with T1D, who have a 15 times higher risk of developing stage 3 T1D compared to the general population. However, since > 85% of people with T1D do not have a family history, general population screening efforts have been started.

There are now several different screening programs in the UK identifying children, young people and adults with IAbs. It is anticipated that there are approximately 700 such children and adults from the different research platforms. These individuals do not typically present to their general practitioner as they have no symptoms, and therefore it is extremely rare to know of such individuals in the UK. Individuals can also be identified from clinical care (personal communication Besser & Randell, BSPED). In order to answer our research questions, the investigators need a mechanism to identify, recruit and consent such individuals into a single combined registry.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 6 months - 70 years
* IAb positive (≥ 1) to any of the following: insulin/GAD/IA2/ZnT8, confirmed in a reference laboratory.
* Participant is willing and able to give informed consent for participation in the study (≥ 16 years old), or for < 16 years, parental/guardian consent (plus assent, where appropriate)
* Living in the UK
* For ADDRESS-2 participants only: have taken part in a blood draw as part of ADDRESS-2
* For the qualitative interviews: Have been living with (or is a parent/guardian of a child who has been living with) a positive IAb result for ≥ 6 months.

Exclusion Criteria:

* Ongoing subcutaneous insulin requirement

Ages: 6 Months to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Potential participants will be identified via:
  * Established research platforms e.g. BOX, INNODIA, ADDRESS-2, PoINT, SINTIA, TrialNet, ELSA, T1DRA, (this is not an exhaustive list)
  * Referral from clinical care
  * Self-referral
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2025-07-11 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Number of individuals enrolled on the registry | 36 months

SECONDARY OUTCOMES:
Participants' perspectives and experiences | 28 months
  Interviews, to to understand the lived experience of being IAb positive or having a child who is IAb positive.
Participants' perspectives and experiences | 28 months
  Interviews, to understand people's information and support needs when living with an IAb result, to improve the information and support given to people and their families who receive a positive T1D IAb result in the future and create a position statement informed by our findings.
Frequency and risk factors (e.g. antibody profile, age) associated with clinical outcomes incident diabetes as defined by start of insulin use and number of DKA episodes | 28 months
  We will undertake data linkage with routinely collected NHS clinical datasets held by NHSE (and the equivalent for the devolved nations)
Frequency and risk factors (e.g. antibody profile, age) associated with HbA1c mmol/l | 28 months
  To undertake data linkage with routinely collected NHS clinical datasets held by NHSE (and the equivalent for the devolved nations)
Frequency of attendance in primary care | 36 months
  To assess the status of being IAb positive on health service usage and clinical outcomes using comparator cohorts (e.g. CPRD/HES)
Frequency of attendance and inpatient admission to secondary/ tertiary care | 36 months
  To assess the status of being IAb positive on health service usage and clinical outcomes using comparator cohorts (e.g. CPRD/HES)
IAb type (IA, IA-2, ZnT8, GAD, ICA) | 36 months
  To compare IAb characteristics to similar cohorts from international registries
IAb laboratory (location) | 36 months
  To compare IAb characteristics to similar cohorts from international registries
IAb titre (mULN) | 36 months
  To compare IAb characteristics to similar cohorts from international registries
Demographic data | 36 months
  To compare demographic characteristics to similar cohorts from international registries
Time to clinical diagnosis (defined as stage 3 T1D) according to standard diagnostic criteria | 36 months
  To assess risk of progression to stage 3 T1D in IAb positive individuals in the UK
Number of individuals who have consented and enrolled to the registry | 36 months
  To assess consent to the registry vs enrolment
IAb number (1-4) | 36 months
  To compare the proportion identified as confirmed positive from clinical care vs reference laboratories
IAb type (IA-2, IA, ZnT8, GAD, ICA) | 36 months
  To compare the proportion identified as confirmed positive from clinical care vs reference laboratories
IAb titre (mULM) | 36 months
  To compare the proportion identified as confirmed positive from clinical care vs reference laboratories

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Besser, Principal Investigator — University of Oxford
Locations (1):
- University of Oxford, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
All IPD will be considered for data sharing.
Supporting Information: Study Protocol, ICF
Time Frame: Access to data will not be considered until after the primary publication for the registry has been published
Access Criteria: Subject to participant consent, data will be shared with other researchers for research projects that have appropriate ethical approval. Requests for access to the data will be controlled by the Data Access Committee.

REFERENCES:
- See also: Related Info — http://www.ukiab.org